CLINICAL TRIAL: NCT07406477
Title: The PROTECT-HIE Trial: Prophylactic Therapy to Enhance Cardiovascular Treatment in Neonatal Hypoxemic Ischemic Encephalopathy
Brief Title: The PROTECT-HIE Trial
Acronym: PROTECT-HIE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Aimann Surak, Principal Investigator, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00162062
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hypoxic-ischemic Encephalopathy (HIE)
Keywords: Hypoxic-ischemic encephalopathy; feasibility RCT; neonatal cardiac dysfunction; prophylactic inotrope; therapeutic hypothermia; neonatal HIE; dobutamine
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Dobutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dobutamine group (Experimental): If randomized to the prophylaxis/dobutamine arm, dobutamine will be administered at a dose of 10 mcg/kg/min via intravenous access within 4 hours of initiating TH. As a part of standard care for HIE, a central umbilical venous access is routinely acquired whenever possible. We will use the dobutamine concentration of 2000 mcg/ml. The infusion will be prepared in dextrose 5% solution in 50 mL bags. Dobutamine monograph is attached to the protocol as well (Appendix F). The infusion will be continued until either weaned by the clinical team, escalation of inotropic support, or improvement of clinical situation to allow weaning of dobutamine.
  Interventions: Drug: Dobutamine; Diagnostic Test: TnECHO
- Control group (Placebo Comparator): Infants randomized to the placebo arm will receive an inert preparation containing no active pharmacologic agent. The placebo will be identical in appearance, volume, and method of administration to the active intervention and will be administered according to the same dosing schedule and duration. We will use dextrose 5% (as placebo), which will be started within 4 hours of initiating TH. The infusion will be continued until either weaned by the clinical team, escalation of inotropic support, or improvement of clinical situation to allow weaning of dobutamine.
  Interventions: Diagnostic Test: TnECHO

INTERVENTIONS:
Drug: Dobutamine — If randomized to the prophylaxis/dobutamine arm, dobutamine will be administered at a dose of 10 mcg/kg/min via intravenous access within 4 hours of initiating TH. As a part of standard care for HIE, a central umbilical venous access is routinely acquired whenever possible. We will use the dobutamine concentration of 2000 mcg/ml. The infusion will be prepared in dextrose 5% solution in 50 mL bags. Dobutamine monograph is attached to the protocol as well (Appendix F). The infusion will be continued until either weaned by the clinical team, escalation of inotropic support, or improvement of clinical situation to allow weaning of dobutamine.
  Arms: Dobutamine group
Diagnostic Test: TnECHO — In both groups, 2 TnECHOs will be performed. TnECHO T1 will be performed within the 24 hours of randomization, and TnECHO T2 will be performed within 24-48 hours after TnECHO T1. All echocardiographic assessments are done by physicians trained in TnECHO or by pediatric cardiology team. Echocardiographic assessment will be performed as per the American Society or Echocardiography guidelines(63-66). Details of the standardised echo views and measurements are outlined in Appendix B.

SUMMARY:
Some babies experience a lack of oxygen and blood flow around the time of birth. This can lead to a serious condition called hypoxic-ischemic encephalopathy (HIE), which can injure the brain and other organs, including the heart. To reduce brain injury, babies with HIE are treated with therapeutic hypothermia, a standard treatment in which the baby's body temperature is carefully lowered for several days. While cooling helps protect the brain, many babies with HIE still develop heart problems and low blood flow, which may worsen outcomes.

Doctors often use medications to support the heart and circulation in these babies, but there is no clear agreement on which medication works best or when it should be started. One commonly used medication is dobutamine, which helps the heart pump more effectively. Dobutamine is already used in newborn intensive care units when babies show signs of heart weakness, but it is usually started only after problems develop.

The PROTECT-HIE trial aims to find out whether it is possible and safe to start dobutamine early, before clear signs of heart failure appear, in newborns with HIE who are receiving therapeutic hypothermia. The idea is that early support of the heart may improve blood flow to vital organs, including the brain, and potentially reduce injury.

In this study, 40 newborns with HIE will take part at a single neonatal intensive care unit. Babies will be randomly assigned to one of two groups. One group will receive a low, preventative dose of dobutamine within the first four hours after cooling begins. The other group will receive a placebo (an inactive fluid that looks the same). Neither the families nor the medical team assessing outcomes will know which treatment the baby received.

The main goal of this study is to determine feasibility-that is, whether starting dobutamine early during cooling can be done reliably and safely in this setting. Researchers will also collect information on important health outcomes, such as signs of brain injury on MRI, seizures, need for additional heart medications, heart function on ultrasound, recovery of blood markers, urine output, length of hospital stay, and survival.

Because HIE is an emergency condition and treatment must start very soon after birth, parents will be approached for consent after the baby has been stabilized. This approach is commonly used in neonatal emergency research and has been approved in similar studies.

The results of this study will help determine whether a larger trial should be done in the future. Ultimately, this research aims to improve care and outcomes for babies affected by HIE by optimizing support for the heart during a critical period after birth.

DETAILED DESCRIPTION:
Purpose

The purpose of this study is to evaluate the feasibility and safety of initiating prophylactic dobutamine infusion in newborns with hypoxic-ischemic encephalopathy (HIE) who are undergoing therapeutic hypothermia (TH). Infants with HIE frequently experience cardiovascular instability during the early postnatal period, which may negatively affect cerebral perfusion and overall outcomes. This study aims to determine whether early, preventive cardiovascular support can be reliably implemented and whether it may be associated with improved short-term clinical outcomes.

Hypothesis

The primary hypothesis is that initiating prophylactic dobutamine infusion within the first four hours of therapeutic hypothermia in newborns with HIE is feasible and safe.

The secondary hypothesis is that early dobutamine prophylaxis may be associated with improved short-term in-hospital outcomes, including reduced severity of brain injury, improved cardiac function, and reduced need for escalation of cardiovascular support.

Justification

HIE remains a major cause of neonatal mortality and long-term neurodevelopmental impairment despite the widespread use of therapeutic hypothermia. Up to 80% of infants with HIE experience some degree of cardiovascular compromise, particularly involving right ventricular dysfunction, which has been associated with worse neurological outcomes and increased mortality.

Although vasoactive medications are frequently used in this population, there is no standardized or evidence-based approach regarding the optimal agent or timing of initiation. Dobutamine is a commonly used inotropic agent in neonates, with a favorable physiological profile that enhances cardiac contractility without significant increases in heart rate or systemic vascular resistance. Preliminary observational data suggest that dobutamine improves cardiac output in infants with HIE undergoing hypothermia.

Currently, dobutamine is typically initiated only after cardiovascular compromise becomes clinically apparent. A prophylactic approach, initiated early during therapeutic hypothermia, may help stabilize cardiac function, optimize systemic and cerebral perfusion, and potentially reduce secondary brain injury. Before a definitive efficacy trial can be conducted, it is necessary to establish the feasibility, safety, and protocol adherence of such an intervention. This pilot randomized controlled trial is designed to address that critical knowledge gap.

Objectives

Primary Objective

To determine the feasibility of initiating prophylactic dobutamine infusion within the first four hours of starting therapeutic hypothermia in newborns with HIE.

Secondary Objectives

To explore whether prophylactic dobutamine is associated with improved short-term clinical outcomes, including:

Presence and severity of brain injury on MRI Mortality Seizure activity (clinical or electrographic) Need for escalation of inotropic or vasoactive support Echocardiographic measures of cardiac function and pulmonary hemodynamics Time to normalization of lactate Duration of inhaled nitric oxide therapy, if required Urine output at 24, 48, and 72 hours Length of hospital stay until discharge or death Research Method / Procedures

This study is a single-center, double-blinded, randomized controlled feasibility trial conducted in a tertiary neonatal intensive care unit.

Eligible participants are newborns diagnosed with hypoxic-ischemic encephalopathy who are receiving therapeutic hypothermia. Infants will be excluded if they have congenital anomalies, contraindications to dobutamine, significant arrhythmias, or if they have already been started on inotropic support prior to randomization.

Participants will be randomized in a 1:1 ratio to either:

Intervention group: Prophylactic dobutamine infusion at 10 mcg/kg/min Control group: Placebo infusion (dextrose 5%) identical in appearance and administration Randomization will be computer-generated, with allocation concealment ensured through a secure REDCap system. The study will be double-blinded; parents, clinical staff, outcome assessors, and data analysts will remain unaware of group assignment until completion of the final analysis.

The assigned infusion (dobutamine or placebo) will be initiated within four hours of starting therapeutic hypothermia and continued until clinical improvement, escalation of cardiovascular support, or weaning at the discretion of the clinical team.

All participants will undergo standardized targeted neonatal echocardiography at two predefined time points during the first 48 hours. Clinical data will be collected throughout hospitalization, including laboratory results, imaging findings, medication use, adverse events, and outcomes.

Due to the emergency nature of HIE and the need for timely initiation of treatment, a deferred consent model will be used. Parents of surviving infants will be approached for written consent as soon as feasible after stabilization and prior to discharge. For infants who die before consent can be obtained, a waiver of consent will be requested for collection of minimal anonymized data.

Plan for Data Analysis

The primary analysis will focus on feasibility outcomes, including:

Proportion of eligible infants successfully receiving the intervention within four hours of initiating therapeutic hypothermia Protocol adherence rate The study will be considered feasible if more than 60% of eligible infants are recruited and more than 75% of randomized infants receive the assigned intervention without major protocol deviations.

Secondary clinical outcomes will be analyzed descriptively, as this pilot study is not powered to detect definitive efficacy differences. Continuous variables will be summarized using means, standard deviations, medians, and interquartile ranges as appropriate. Categorical variables will be reported as frequencies and percentages.

Comparisons between groups will be conducted using:

Student's t-test or Mann-Whitney U test for continuous variables Chi-square test for categorical variables All analyses will follow the intention-to-treat principle. Statistical significance will be defined as a two-sided p-value <0.05. Analyses will be performed using IBM SPSS and SAS statistical software after database lock and unblinding.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with hypoxemic ischemic encephalopathy (HIE) receiving therapeutic hypothermia (TH).

Exclusion Criteria:

1. Congenital abnormality
2. known contraindication of dobutamine

   * Left ventricular outflow tract dynamic obstruction
   * Hypersensitivity to dobutamine
   * Uncorrected tachyarrhythmias or ventricular fibrillation
3. Newborns who are already started on inotropes at the time of randomization.
4. Parental refusal to consent to participate

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility/Safety | At 24 hours of age
  Proportion of eligible infants receiving the intervention (or placebo) within 4 hours of initiating TH

SECONDARY OUTCOMES:
Short term outcomes | through study completion, an average of 1 month
  Brain injury on MRI (normal/abnormal)
Short term outcomes | through study completion, an average of 1 month
  Severity and type of brain injury [as per reference # 72 in the uploaded protocol, Mohammad K, et al. Consensus Approach for Standardization of the Timin]
Short term outcomes | through study completion, an average of 1 month
  Death (yes/no)
Short term outcomes | through study completion, an average of 1 month
  Presence of seizure activity (clinical or electrical) (yes/no)
Short term outcomes | through study completion, an average of 1 month
  Need for escalation the inotropic support (beyond the above-mentioned infusions) (yes/no)
Short term outcomes | through study completion, an average of 1 month
  Echocardiographic parameters (TAPSE in mm, RV FAC in %, LV EF in %)
Short term outcomes | through study completion, an average of 1 month
  - Time to normalizing lactate reported in hours (the cutoff for normal lactate is 3 as per local laboratory values)
Short term outcomes | through study completion, an average of 1 month
  Duration of inhaled nitric oxide if needed reported in hours (from the time of initiation to time of discontinuation)
Short term outcomes | through study completion, an average of 1 month
  Urine output at 24, 48, and 72 hours reported in cc/k/hour
Short term outcomes | through study completion, an average of 1 month
  Length of stay in hospital till discharge in days (defined from the date of birth till the date of discharge/death)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided